CLINICAL TRIAL: NCT01548027
Title: Efficacy of Surgical Transversus Abdominis Plane Block for Postoperative Pain Relief Following Abdominal Surgery in Pediatric Patients.
Brief Title: Surgical Transversus Abdominis Plane Block in Pediatric Patients
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 752/2554
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Child
Keywords: TAP block; postoperative analgesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No intervention (Experimental): no injection of local anesthetic agents
  Interventions: Other: No intervention
- Local infiltration group (Experimental): patients would have 0.5 ml/kg of 0.25% bupivacaine if age < 6 months or 1 ml/kg if age > 6 months around the wound by surgeon. The needle will be injected in subcutaneous tissue parallel to the wound.
  Interventions: Procedure: Local infiltration group
- TAP block group (Experimental): Surgical TAP block (sTAP: Patients would have 0.5 ml/kg of 0.25% bupivacaine if age < 6 months or 1 ml/kg if age > 6 months
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: Local infiltration group — patients would have 0.5 ml/kg of 0.25% bupivacaine if age < 6 months or 1 ml/kg if age > 6 months around the wound by surgeon. The needle will be injected in subcutaneous tissue parallel to the wound.
  Other Names: local anesthetic infiltration
  Arms: Local infiltration group
Procedure: TAP block — Surgical TAP block (sTAP: Patients would have 0.5 ml/kg of 0.25% bupivacaine if age < 6 months or 1 ml/kg if age > 6 months
  Other Names: surgical transversus abdominis plane block
  Arms: TAP block group
Other: No intervention — No intervention
  Arms: No intervention

SUMMARY:
The objective of this study to determine the effect of surgical transversus abdominis plane block and local infiltration for postoperative pain control in major abdominal surgery compare with control group.

DETAILED DESCRIPTION:
Most children experience postoperative pain after major abdominal surgery. They may have ineffective ventilation, following atelectasis and pneumonia if receive inadequate pain management. There are several methods used for pain relief such as epidural block, intravenous analgesia with local infiltration, transversus abdominis plane (TAP) block by ultrasound guided and surgical TAP block. Therefore, the investigators would like to compare the effectiveness of postoperative pain control with TAP block. However, TAP block in children need experience and ultrasound. The investigators decided to do surgical TAP block performing by inject from peritoneum point to skin instead.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 15 year
2. ASA I-III
3. Abdominal surgery : all upper abdomen and lower abdomen which would have midline incision
4. Elective surgery

Exclusion Criteria:

1. Allergic to Lidocaine or bupivacaine
2. Delayed development
3. Major abdominal surgery within 2 year

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
opioids consumption | 24 hours
  total opioids consumption in first 24 hours postoperatively

SECONDARY OUTCOMES:
Time to first analgesic | 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Saowaphak Lapmahapaisan, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand